CLINICAL TRIAL: NCT05491967
Title: Comparison of Vascular Risk in Patients Treated for Obstructive Sleep Apnea/Hypopnea Syndrome (OSAHS) With Continuous Positive Airway Pressure (CPAP) and Mandibular Advancement Orthosis
Brief Title: Comparison of Vascular Risk in Patients Treated for Obstructive Sleep Apnea/Hypopnea Syndrome
Acronym: SAHOSVAS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Valence (Other)
Responsible Party: Sponsor
Other Study IDs: RIPH-CHV-07
Record Dates: First submitted 2022-07-08; First posted 2022-08-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Obstructive Sleep Apnea/Hypopnea Syndrome
Keywords: cardiovascular risk
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Continuous Positive Airway Pressure (CPAP): Obstructive Sleep Apnea/Hypopnea Syndrome treated with Continuous Positive Airway Pressure (CPAP
- Mandibular Advancement Orthosis: Obstructive Sleep Apnea/Hypopnea Syndrome treated with Mandibular Advancement Orthosis

SUMMARY:
a monocentric,non interventional, prospective study to compare cardiovascular risk in patients with Obstructive Sleep Apnea/Hypopnea Syndrome treated with Continuous Positive Airway Pressure (CPAP) and Mandibular Advancement Orthosis.

DETAILED DESCRIPTION:
The first-line treatment of severe Obstructive Sleep Apnea/Hypopnea Syndrome (OSAHS) is nocturnal ventilation with Continuous Positive Airway Pressure (CPAP). and The second-line treatment is the mandibular advancement orthosis (MAO)].

CPAP is the most effective treatment to reduce the apnea-hypopnea index (AHI). However, its tolerance is sometimes difficult, causing many discontinuations.

The purpose of this review is to evaluate a vascular morbimortality criteria:

* Cardiovascular: myocardial infarction, heart failure, rhythm disorder
* Neurological: transient or non transient stroke
* ophthalmologic: anterior ischemic optic neuropathy, occlusion of the central artery or central retinal vein occlusion

ELIGIBILITY:
Inclusion Criteria:

* Obstructive Sleep Apnea/Hypopnea Syndrome treated with With Continuous Positive Airway Pressure (CPAP) or Mandibular Advancement Orthosis
* Age ≥ 18 years old
* Read, write and understand the French language

Exclusion Criteria:

* Patient under guardianship, deprived of liberty, safeguard of justice
* Refusal to participate in research

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Obstructive Sleep Apnea/Hypopnea Syndrome treated with With Continuous Positive Airway Pressure (CPAP) or Mandibular Advancement Orthosis
Sampling Method: Non-Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2023-03-16 (Actual)

PRIMARY OUTCOMES:
morbimortality vascular criteria | up to 6 months
  Presence or absence of cardiovascular event
morbimortality vascular criteria | up to 6 months
  Presence or absence of neurologic event
morbimortality vascular criteria | up to 6 months
  Presence or absence of ophthalmologic event

CONTACTS AND LOCATIONS:
Locations (1):
- Ch Valence, Valence, Drome, France